CLINICAL TRIAL: NCT06135441
Title: Bone Manifestation of Nutritional Disorders Among Infants and Pre-school Children Attending Assiut University Children Hospital
Brief Title: Bone Manifestation of Nutritional Disorders Among Infants and Pre-school Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eslam Hamam Ebrahim, Principal Investigator, Assiut University
Other Study IDs: Bone manifestation
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Bone Loss; Nutrition Disorders
MeSH Terms: conditions — Bone Diseases, Metabolic; Nutrition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Nutrients important to bones. Because bones undergo continuous remodeling, an adequate supply of nutrient substrate is needed to support the formation phase of bone remodeling. In addition to their passive roles as substrate for bone formation, dietary calcium and protein play active roles in bone metabolism, as well as phosphorus and vitamin D. Other vitamins and minerals are also needed for metabolic processes related to bone, directly or indirectly.

DETAILED DESCRIPTION:
Nutrients important to bones. Because bones undergo continuous remodeling, an adequate supply of nutrient substrate is needed to support the formation phase of bone remodeling. In addition to their passive roles as substrate for bone formation, dietary calcium and protein play active roles in bone metabolism, as well as phosphorus and vitamin D. Other vitamins and minerals are also needed for metabolic processes related to bone, directly or indirectly.

The Food and Nutrition Board (FNB) of the National Academy of Sciences, has released in the past few years the new Dietary Reference Intakes (DRI) based on the latest understanding about nutrient requirements for optimizing health.

The fetal period, early life, childhood, and puberty are critical periods for the development and/or programming of metabolic systems, including the skeleton. Osteoporosis is described by the World Health Organization (WHO) as a progressive systemic skeletal disease characterized by low bone mass and microarchitectural deterioration of bone tissue, with a consequent increase in bone fragility and susceptibility to fracture. Because of the morbidity of osteoporosis, the prevention of this disease and its associated fractures is considered essential to the maintenance of health, quality of life, and independence in the elderly population.

Peak bone mass attained during childhood and adolescence determines skeletal fragility in old age.

Peak bone mass is the amount of bone acquired when accrual ceases or reaches a plateau at some point after the completion of growth and development. Metabolic bone disease (MBD) is an umbrella term that encompasses a broad spectrum of clinically different diseases that share the common finding of an aberrant bone chemical milieu leading to a defective skeleton and bone abnormalities. Metabolic bone diseases are usually characterized by a dramatic clinical presentation and manifestation that are commonly reversible once the underlying defect has been treated. Abnormalities of minerals include calcium, phosphorus, magnesium, or vitamin D developing as a result of dysfunctions of the various factors that control mineral homeostasis. The defective mineralization translates into rickets at the level of the epiphyseal growth plates and osteomalacia on the endocortical and cancellous bone surfaces Moreover, osteogenesis imperfecta (OI) pathogenesis has been expanded from a simple collagen defect to abnormalities in bone cell metabolism and development with primary defects in osteoblast differentiation. Metabolic bone disease is to be differentiated from skeletal dysplasia which are a larger group of genetic bone disorders that overlaps with MBD. In contrast to MBD, skeletal dysplasias are heritable diseases that have generalized abnormalities in cartilage and bone. The primary defects are in specific signal system or cell types that orchestrate processes of skeleton formation causing the bone disorder.

ELIGIBILITY:
Inclusion Criteria:

* All malnutrition cases attending the nutrition out-patient clinic in AUH

Exclusion Criteria:

* bone disorders in non-malnourished cases
* bone disease due to a genetic disorder

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children from month till age of 18 years attending to Assiut university children hospital's metabolic, nutrition and orthopedic clinics with short statue, bone deformity or anomaly.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of bone affection by nutritional disorders in Assiut University Hospital. | Baseline
  The prevalence of bone affection by nutritional disorders in Assiut University Hospital.
Different manifestations of bone affection by nutritional disorders | Baseline
  Different manifestations of bone affection by nutritional disorders